CLINICAL TRIAL: NCT06069947
Title: Sequential Adult Left Lateral Lobe Liver Transplantation (SALT) in Patients With Liver Cirrhosis With Hepatocellular Carcinoma(HCC): a Single-center, Prospective, Single-arm Study
Brief Title: SALT for Liver Cirrhosis With HCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-185-C
Record Dates: First submitted 2023-09-22; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: HCC; Liver Cirrhosis
Keywords: Hepatocellular Carcinoma; Liver cirrhosis; Liver transplantation; Two-stage liver resection
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: SALT operation plan for patients who meet the enrollment conditions and successfully match the donor liver: Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical group (Experimental): SALT operation plan for patients who meet the enrollment conditions and successfully match the donor liver: Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.
  Interventions: Procedure: sequential adult left lateral lobe liver transplantation (SALT)

INTERVENTIONS:
Procedure: sequential adult left lateral lobe liver transplantation (SALT) — Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.

SUMMARY:
HCC is the third leading cause of cancer deaths worldwide. Although surgical treatment may be effective in patients with HCC, the five-year survival rate is only 50-70%. Moreover, due to the lack of early diagnostic marker, most patients with HCC are often diagnosed in an advanced stage with poor prognosis. Therefore, there is an urgent need to further understand the possible aetiological factors and surgical treatment methods to improve the prognosis of patients with HCC. Liver transplantation is an ideal choice for patients with liver cirrhosis with HCC, which can significantly improve the postoperative survival rate. But the most serious problem facing such patients is the shortage of donor livers. In 2015, Norwegian scholars proposed a new surgical method, that is, resection and partial liver segment (2-3 segment) transplantation combined with delayed total hepatectomy can greatly alleviate the shortage of liver donors in the above-mentioned patients. Based on the experience of clinical operation, our center proposes and designs a clinical study of sequential adult left lateral lobe liver transplantation (SALT) for the treatment of patients with liver cirrhosis with HCC. On the basis of RAPID, the safety and efficacy of sequential adult left lateral lobe liver transplantation were evaluated for the above patients.

DETAILED DESCRIPTION:
Heoatocellular carcinoma (HCC) ranks sixth in the incidence of malignant tumors and fourth in case fatality in the world. In China, liver cancer deaths account for the second largest cause of all cancer deaths. Surgical resection of liver cancer is still the main treatment, but the five-year survival rate is only 50%-70%. Liver transplantation can remove tumours and the underlying liver disease at the same time, and has become an important means for the radical treatment of liver cancer.

Liver transplantation for liver cancer is a tortuous process. The original intention of liver transplantation was to treat "unresectable liver cancer", but due to the high recurrence rate and metastasis rate of postoperative tumors, many centers list liver cancer as a contraindication to liver transplantation. In 1996, Mazzaferro et al. proposed the Milan criteria, and patients with liver cancer patients has a 4-year survival rate of 85% after liver transplantation. However, the Milan criteria was too strict and excluded a large number of patients with liver cancer who were likely to survive for a long time through liver transplantation. Therefore, the UCSF standard was proposed in 2001, and the small relaxation was made on the basis of the Milan criteria, and the survival rate was similar to the Milan criteria. In China, hepatitis B virus infection accounts for the vast majority of liver cancer patients, and the race, liver cancer incidence and treatment concept are different from European and American countries, and many factors indicate that it is urgent to formulate liver transplantation criteria that meet China's national conditions. In 2006, the Shanghai Fudan criteria was proposed based on the clinical data of liver transplant patients in China, which further expanded the scope of indications for liver transplantation of liver cancer, and did not reduce the overall survival rate and tumor-free survival rate of patients after surgery, and was also verified in the Western population. Since then, Kyoto standards, Hangzhou standards, Up-To Seven standards, and Toronto standards have been proposed around the world. These criteria have been relaxed to varying degrees in the size and number of tumors. At present, except for the Milan criteria and UCSF criteria, other standards have not been uniformly recognized.

However, it is difficult for patients with cirrhosis with hepatocellular carcinoma (cHCC) to enroll in the above transplant criteria, and many patients lose the opportunity to obtain liver transplantation, so the biggest problem faced by patients with cirrhosis and hepatocellular carcinoma is the shortage of donor liver. Also, cirrhosis with hepatocellular carcinoma is often considered a contraindication to liver transplantation, making it more difficult to obtain a donor liver.

Therefore, expanding the donor liver pool is urgently needed for the treatment of patients with patients with liver cirrhosis with HCC. In 2015, Norwegian scholars proposed a new surgical method, that is, resection and partial liver segment 2-3 transplantation with delayed total hepatectomy (RAPID) . This approach allows transplantation of the left liver (segments 2+3) to an adult recipient, while the remaining enlarged right hemi-liver is transplanted to another adult recipient, effectively avoiding some unsuitable left lateral lobe livers for pediatric recipients to be wasted. Recipients who received right-hemi-liver transplantation had a similar prognosis compared with those who received whole-liver transplantation. Therefore, if the RAPID technique is confirmed to be feasible, it can greatly alleviate the shortage of liver donors. In addition to cadaver sources, living adult donors can also be considered as the source of liver donors. A smaller left lateral lobe donor liver also places less burden on the donor than a left or right hemiliver.

To sum up, our center proposed and designed a clinical study of sequential adult left lateral lobe liver transplantation (SALT) in the treatment of patients with liver cirrhosis with HCC based on clinical surgical experience. On the basis of RAPID surgery, the overall survival rate of patients with liver cirrhosis with HCC was evaluated by SALT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75;
2. Child-Pugh A-B ;
3. liver cirrhosis with Heoatocellular Carcinoma (HCC) with Hepatitis B virus infection 4. Patients with Heoatocellular Carcinoma (HCC) meets the "up to seven" criteria: the sum of tumour size and tumour numbers does not exceed 7;

5. Performance Status 0-1; 6. Sign the informed consent form.

Exclusion Criteria:

1. Combined with the main portal vein tumor thrombus, the main vena cava tumor thrombus and common bile duct tumor thrombus;
2. Combined with severe hepatic encephalopathy ;
3. Combined with pulmonary hypertension(high-risk or middle-risk, WHO grade: III-IV);
4. Special types of anatomical variations(such as portal vein classification: type III and type IV, etc. );
5. Extrahepatic tumor burden;
6. Cardiopulmonary disease or severe infection or Cerebral Vascular Disease that cannot be corrected, with high surgical risk, that makes liver transplantation impossible;
7. Psychological or social conditions may interfere with the patient's participation in the study or evaluation of the study results;
8. Other reasons that the researchers think are not suitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 3 years after the second liver resection
  To describe overall survival in patients with liver cirrhosis with HCC treated with sequential adult left lateral lobe liver transplantation.

SECONDARY OUTCOMES:
Disease-free survival，DFS | 1 month, 3 months, 6 months, 1 year, 2 years and 3 years post-transplant
  Describe the tumor-free survival period of SALT in the treatment of patients with liver cirrhosis with HCC

IPD SHARING:
Plan to Share IPD: No